CLINICAL TRIAL: NCT04075136
Title: OCTA-Directed PDT Triple Therapy for Treatment-Naïve Patients With Exudative Age-Related Macular Degeneration Versus Standard of Care Anti-VEGF(Anti-vascular Endothelial Growth Factor) Monotherapy
Brief Title: Optical Coherence Tomography Angiography (OCTA) - Directed PDT Triple Therapy
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: IRB stopped study due to safety concerns before any participants were enrolled.
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Modulight (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00058375
Record Dates: First submitted 2019-08-29; First posted 2019-08-30 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2023-04

CONDITIONS: Exudative Age Related Macular Degeneration
Keywords: Macular degeneration; Lucentis; Triescense; Photodynamic laser treatment
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab; Triamcinolone Acetonide; Triamcinolone; Verteporfin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (3):
- Arm A: Lucentis (Active Comparator): A standard of care treatment of 0.05ml/0.5mg Lucentis given every 4 weeks for 48 weeks.
  Interventions: Drug: Ranibizumab
- Arm B: Lucentis & PDT Laser (Experimental): A one time treatment of 0.05ml/0.5mg Lucentis in combination with PDT laser administered at half-fluence.
  Interventions: Drug: Ranibizumab; Device: Photodynamic laser treatment (PDT); Drug: verteporfin
- Arm C: Lucentis, PDT Laser and Triescense (Experimental): A one time treatment of 0.05ml/0.5mg Lucentis in combination with PDT laser administered at half-fluence and an intravitreal injection of 0.5ml-2mg Triescence at the time of PDT treatment.
  Interventions: Drug: Ranibizumab; Device: Photodynamic laser treatment (PDT); Drug: Triamcinolone Acetonide; Drug: verteporfin

INTERVENTIONS:
Drug: Ranibizumab — Intravitreal injection 0.5 MG Per 0.05 ML Injection.
  Other Names: Lucentis
Device: Photodynamic laser treatment (PDT) — PDT light dose of 50 J/cm2 of neovascular lesion administered at an intensity of 600mW/cm2. A Visudyne infusion will be administered for the PDT portion of the treatment at a dose of 6mg/m2 body surface area. PDT will be administered at half-fluence - measured by time, i.e. 42 seconds as opposed to full-fluence which is 83 seconds.
  Arms: Arm B: Lucentis & PDT Laser; Arm C: Lucentis, PDT Laser and Triescense
Drug: Triamcinolone Acetonide — Intravitreal injection of 0.5ml-2mg
  Other Names: Triesence
  Arms: Arm C: Lucentis, PDT Laser and Triescense
Drug: verteporfin — Visudyne infusion will be administered for the PDT portion of the treatment at a dose of 6mg/m2 body surface area.
  Other Names: Visudyne
  Arms: Arm B: Lucentis & PDT Laser; Arm C: Lucentis, PDT Laser and Triescense

SUMMARY:
Optical Coherent Tomography Angiography (OCTA)-Directed PDT Triple Therapy for Treatment-Naïve Patients with Exudative Age-related Macular Degeneration (ARMD) versus Standard of Care Anti-VEGF Monotherapy

DETAILED DESCRIPTION:
This study is a 48 week, single center, randomized controlled clinical trial. Approximately 150 subjects will be randomized into three separate arms. This study compares the efficacy of standard of care Lucentis (ranibizumab) monotherapy versus OCTA-Directed PDT Triple Therapy with Lucentis (ranibizumab), PDT with Visudyne (verteporfin), and Triescence (triamcinolone acetonide) in treatment-naïve patients with Exudative Age-Related Macular Degeneration. OCTA-Directed PDT Double Therapy with Lucentis (ranibizumab) and PDT with Visudyne (verteporfin) will also be tested to confirm the hypothesis that steroids are necessary.

ELIGIBILITY:
Inclusion Criteria:

* Willing to give written informed consent
* Willing and able to comply with all study procedures for the duration of the study.
* Presence of Exudative ARMD with evidence of choroidal neovascularization: type 1, 2, and/or 3 on spectral domain OCT, fluorescein angiography, indocyanine green angiogram and optical coherent tomography angiography
* Visual Acuity of 20/25 to 20/400 at screening and baseline visits using an autorefractor or Early Treatment Diabetic Retinopathy Study
* Intraocular pressure less than or equal to 25mmHG
* Females of childbearing potential that are willing to use medically acceptable methods of birth control.

Exclusion Criteria:

* Exudation maculopathies without drusen
* Previous treatment with macular photocoagulation, anti-VEGF medication or PDT with Visudyne
* Myocardial infarction or cerebrovascular accident within the last 6 weeks
* Previous vitrectomy
* Optic neuropathy
* Diabetic retinopathy
* Traction maculopathies
* Allergies to fluorescein and indocyanine, dilating agents or anti-VEGF medications
* Have received previous treatment for ARMD
* Any uncontrolled condition or illness that in the opinion of the investigator makes the subject unsuitable for the study

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-03-30 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of subretinal exudation resolution | 6 months
  The percentage of subretinal exudation resolution
Percentage of intraretinal exudation resolution | 6 months
  The percentage of intraretinal exudation resolution

SECONDARY OUTCOMES:
Percentage of subretinal exudation resolution | 12 months
  Subretinal exudation resolution
Percentage of intraretinal exudation resolution | 12 months
  Intraretinal exudation resolution
Best corrected visual acuity (BCVA) | Baseline
  Best corrected visual acuity
Best corrected visual acuity (BCVA) | 12 months
  Best corrected visual acuity
Duration of treatment effect | Up to 6 months
  Duration of treatment effect
Foveal thickness | Baseline
  Measured using Optical coherence tomography (OCT)
Foveal thickness | 12 Months
  Measured using Optical coherence tomography (OCT)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Nelson, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Results will updated once final analysis is complete.